CLINICAL TRIAL: NCT00454103
Title: Evaluation of 123I-Iodometomidate for Adrenal Scintigraphy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wue_123IMTO_100/05
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2007-10

CONDITIONS: Adrenal Tumor; Adrenocortical Carcinoma
Keywords: adrenocortical carcinoma (ACC); adrenal tumor; metastastic adrenocortical carcinoma
MeSH Terms: conditions — Adrenal Gland Neoplasms; Adrenocortical Carcinoma | interventions — iodophenyl metomidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 123I-Iodometomidate

SUMMARY:
The improvement of conventional imaging techniques has led to an increased detection rate of different adrenal tumors. Since those tumors can belong to a variety of entities the therapeutic consequences also show considerable variation. In order to definitely determine the type of tumor, invasive procedures like CT guided biopsies are often required, which could be avoided by a tumor specific imaging method. The presently available scintigraphic procedures are either time consuming and lead to high radiation exposure or are technically demanding. The steroidogenic enzymes CYP11B1 (11ß-hydroxylase)and CYP11B2 (aldosterone synthase)are expressed exclusively in the adrenal cortex and therefore represent suitable targets for a specific imaging technique. In our project we evaluate 123I-Iodometomidate which binds to both CYP11B enzymes as radiotracer for adrenal scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

1. Adrenal tumor seen by CT or MRT-scan with diameter of at least 2 cm or patient with adrenocortical carcinoma and suspected metastasis or local recurrence or patients with primary hyperaldosteronismus and adrenal tumour > 1 cm
2. Hormonal work up of of the adrenal tumor according to ENS@T (European network for the study of adrenal tumours)-criteria
3. Age ≥ 30 Jahre
4. Effective contraception (pearl index <1%)
5. Written informed consent

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Renal insufficiency (serum creatinine > 2,0 mg/dl or MDRD < 60 ml/min)
3. Known allergy to etomidate or constituents of the test drug

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Reiners, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- Würzburg, Germany